CLINICAL TRIAL: NCT07134361
Title: Clinical Analysis and Ultrasound Evaluation of the Median Nerve Cross-sectional Area Before and After Carpal Tunnel Release
Brief Title: Evaluation by Clinical and Hand Ultrasound in Carpal Tunnel Syndrome
Acronym: ECHO-CTS
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcelo Rosa de Rezende, MD, PHD, University of Sao Paulo General Hospital
Other Study IDs: 86571525.4.0000.0068
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome (CTS); Carpal Tunnel Surgery
Keywords: carpal tunnel syndromes; Median Neuropathy; Ultrasonography
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Patients diagnosed with primary carpal tunnel syndrome (CTS) are undergoing open carpal tunnel release as part of their routine clinical care. The surgical procedure is not assigned by the study but performed according to standard practice. The cohort will be followed prospectively with clinical assessments (Boston Carpal Tunnel Questionnaire, QuickDASH, grip and pinch strength, Semmes-Weinstein monofilament testing), as well as ultrasonographic evaluation of the median nerve cross-sectional area, before and at three and six months after surgery, to identify prognostic factors associated with functional and symptomatic recovery.
  Interventions: Procedure: Open Carpal Tunnel Release

INTERVENTIONS:
Procedure: Open Carpal Tunnel Release — All patients included in the cohort will undergo open carpal tunnel release as part of routine clinical care. The study does not assign the surgical procedure as an investigational intervention; however, it will observe clinical and ultrasonographic outcomes before and after surgery to assess prognostic factors.

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a common condition where pressure on the median nerve in the wrist causes pain, numbness, and weakness in the hand. Surgery to release the carpal tunnel is often performed to relieve these symptoms.

This study will evaluate the changes in the median nerve after surgery and how these changes relate to symptom improvement. Investigators will use ultrasound imaging to measure the nerve size before and at three and six months after surgery. Patients will also complete questionnaires about their symptoms and hand function, and undergo tests to assess strength and sensation.

The investigator's goal is to determine whether changes observed on ultrasound are associated with the rate of patient recovery. This may help doctors better monitor healing and improve care for people with CTS.

DETAILED DESCRIPTION:
This is a prospective observational cohort study designed to evaluate structural and functional recovery in patients with primary carpal tunnel syndrome undergoing open carpal tunnel release. The study also aims to identify prognostic factors associated with clinical and functional improvement after surgery. Patients will be consecutively recruited from the Hand Surgery and Microsurgery Department of a tertiary University Hospital.

All participants will undergo a standardized surgical procedure performed by experienced hand surgeons as part of routine clinical care. Ultrasonographic assessments of the median nerve cross-sectional area (CSA) at the carpal tunnel inlet and outlet will be conducted by an experienced radiologist using a high-resolution linear transducer (7-16 MHz) at three time points: preoperatively, and at 3 and 6 months after surgery. Secondary outcomes, including the Boston Carpal Tunnel Questionnaire (BCTQ), QuickDASH, quantitative grip and pinch strength measured with calibrated dynamometers, and tactile sensibility testing with Semmes-Weinstein monofilaments, will be assessed at the same time points by an occupational therapist specializing in hand therapy. This evaluation schedule is designed to characterize both morphological and functional recovery after surgery longitudinally.

The primary outcome is the change in median nerve CSA between baseline and follow-up. Secondary outcomes include changes in BCTQ and QuickDASH scores, grip strength, pinch strength, and sensory thresholds. All analyses will be two-sided with an alpha level of 0.05 and 95% confidence intervals. Data normality will be assessed with the Shapiro-Wilk test. Continuous outcomes will be compared pre- and postoperatively using paired t-tests or Wilcoxon signed-rank tests, as appropriate. Associations between CSA change and secondary outcomes will be examined with univariate and multivariable linear regression, adjusting for age, sex, symptom duration, and dominant hand involvement, with interaction terms to assess potential effect modification. Exploratory subgroup analyses for age, sex, and symptom duration will follow the same statistical approach, and categorical variables, if applicable, will be compared using Chi-square or Fisher's exact tests.

The prognostic value of baseline CSA will be explored using receiver operating characteristic (ROC) curve analysis for clinically meaningful improvement in secondary outcomes at 3 and 6 months. The Youden index will determine the optimal cutoff, and the area under the curve (AUC) will quantify discriminative ability. This cutoff will then stratify patients for exploratory comparisons over time. The sample size was calculated for a paired comparison of pre- and postoperative CSA, assuming a mean detectable difference of 1.0 mm² and a standard deviation of paired differences of 3.29 mm², with an alpha level of 0.05 and 80% power. This yields a requirement of 85 patients; allowing for 20% missingness, the final target is 107 participants.

All analyses will be performed using MedCalc version 23.2.7 (64-bit). Standardized protocols will be applied for all assessments, with regular data validation, source-data verification against medical records, and maintenance of a detailed data dictionary. Standard Operating Procedures will guide recruitment, data collection, and management. Missing data will be addressed using appropriate statistical methods such as multiple imputation or sensitivity analyses, depending on the mechanism and extent of missingness. No experimental interventions will be introduced; the study is observational in nature. Results will contribute to improved understanding of prognostic indicators in carpal tunnel syndrome and support evidence-based postoperative monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary carpal tunnel syndrome (CTS), confirmed by characteristic symptoms, physical examination findings, and a cross-sectional area superior to 10 mm² in the ultrasonography baseline.
* Indication for open carpal tunnel release as part of routine clinical care.

Exclusion Criteria:

* Secondary CTS due to inflammatory arthritis, prior wrist trauma, or space-occupying lesions.
* History of previous carpal tunnel release in the affected hand.
* Concomitant peripheral neuropathies (e.g., diabetic polyneuropathy) or cervical radiculopathy
* Inability to undergo ultrasound assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients referred to the Hand Surgery and Microsurgery Department at Hospital das Clínicas, a tertiary care academic hospital affiliated with the University of São Paulo Medical School in São Paulo, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in median nerve cross-sectional area (CSA) measured by high-resolution ultrasound | Baseline (preoperative) and at 3 and 6 months post-surgery
  The CSA of the median nerve will be assessed at two standardized locations: the carpal tunnel inlet and the carpal tunnel outlet. Measurements will be obtained using a high-frequency linear transducer (7-16 MHz) with the patient seated, forearm resting, and wrist in neutral position. The CSA will be calculated by manually tracing the inner border of the epineurium on transverse images. Assessments will be performed preoperatively and at three and six months postoperatively. The aim is to evaluate structural changes in the median nerve after carpal tunnel release and correlate them with clinical recovery.

SECONDARY OUTCOMES:
Change in Boston Carpal Tunnel Questionnaire (BCTQ) scores | Baseline (preoperative) and at 3 and 6 months post-surgery
  The Boston Carpal Tunnel Questionnaire will be used to assess symptom severity (BCTQ-S) and functional status (BCTQ-F). Each subscale score ranges from 1 (no symptoms or limitations) to 5 (severe symptoms or limitations). Scores will be calculated as the mean of items in each subscale.
Change in QuickDASH scores | Baseline (preoperative) and at 3 and 6 months post-surgery
  The Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire measures upper limb disability and symptoms. Scores range from 0 (no disability) to 100 (most severe disability).
Change in grip and pinch strength | Baseline (preoperative) and at 3 and 6 months post-surgery
  Grip and pinch strength will be measured using a calibrated hand dynamometer and pinch gauge, respectively. Tests will be performed with the participant seated, with the shoulder adducted, the elbow at 90°, and the forearm in a neutral position. The highest value from the three trials will be recorded for each hand.
Change in tactile sensitivity using Semmes-Weinstein monofilaments. | Baseline (preoperative) and at 3 and 6 months post-surgery
  Sensory function will be evaluated using Semmes-Weinstein monofilaments applied to median nerve-innervated areas of the hand. Threshold levels will be classified according to standard color coding (green to red).

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Rosa Rezende, MD, PhD,, Principal Investigator — HOSPITAL DAS CLÍNICAS DA FACULDADE DE MEDICINA DA UNIVERSIDADE DE SÃO PAULO (HCFM/USP)
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the publication (after de-identification) will be shared. This includes clinical and ultrasonographic data collected before and after surgery. Supporting documents such as the study protocol, statistical analysis plan, and analytic code will also be available upon request. Data sharing will comply with ethical approvals and patient consent requirements.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 12 months after publication of the primary results and available for 3 years.
Access Criteria: Data will be made available to researchers whose proposed use of the data has been approved by an independent review committee (data access committee). Access requests should include a methodologically sound proposal and will be evaluated for scientific merit and ethical compliance.
URL: https://zenodo.org/

REFERENCES:
- [Background] Tajika T, Kuboi T, Endo F, Chikuda H. Relationship Between Morphological Change of Median Nerve and Clinical Outcome Before and After Open Carpal Tunnel Release: Ultrasonographic 1-Year Follow-up After Operation. Hand (N Y). 2022 May;17(3):534-539. doi: 10.1177/1558944720937367. Epub 2020 Jul 9. PMID 32643958
- [Background] Jansen MC, Duraku LS, Hundepool CA, Power DM, Rajaratnam V, Selles RW, Zuidam JM. Management of Recurrent Carpal Tunnel Syndrome: Systematic Review and Meta-Analysis. J Hand Surg Am. 2022 Apr;47(4):388.e1-388.e19. doi: 10.1016/j.jhsa.2021.05.007. Epub 2021 Aug 3. PMID 34353640
- [Background] Cavalcante MC, Moraes VY, Oses GL, Nakachima LR, Belloti JC. Quality analysis of prior systematic reviews of carpal tunnel syndrome: an overview of the literature. Sao Paulo Med J. 2022 Dec 19;141(5):e20211020. doi: 10.1590/1516-3180.2021.1020.R2.10102022. eCollection 2022. PMID 36541951
- [Background] Katz JN, Larson MG, Sabra A, Krarup C, Stirrat CR, Sethi R, Eaton HM, Fossel AH, Liang MH. The carpal tunnel syndrome: diagnostic utility of the history and physical examination findings. Ann Intern Med. 1990 Mar 1;112(5):321-7. doi: 10.7326/0003-4819-112-5-321. PMID 2306060
- [Background] Kim JK, Koh YD, Kim JO, Choi SW. Changes in Clinical Symptoms, Functions, and the Median Nerve Cross-Sectional Area at the Carpal Tunnel Inlet after Open Carpal Tunnel Release. Clin Orthop Surg. 2016 Sep;8(3):298-302. doi: 10.4055/cios.2016.8.3.298. Epub 2016 Aug 10. PMID 27583113